CLINICAL TRIAL: NCT05656716
Title: Effect of a Multimodal Intervention on the Response to Neoadjuvant Therapy in Breast Cancer Patients.
Brief Title: Multimodal Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Lucas Jurado-Fasoli, Dr., Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Multimodal Project
Record Dates: First submitted 2022-11-27; First posted 2022-12-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to receive the multimodal intervention (nutrition and exercise)
  Interventions: Behavioral: Nutritional intervention; Behavioral: Physical exercise intervention
- Control group (No Intervention): Participants will not receive the multimodal intervention.

INTERVENTIONS:
Behavioral: Nutritional intervention — The nutritional intervention will be based on a nutritional education program adapted for patients with breast cancer in active treatment. The nutritional intervention program will be based on the practical guidelines for nutrition in the oncology patient. The main objectives of the nutritional intervention will focus on preventing malnutrition, maintaining an adequate nutritional status and dietary adaptation to secondary symptomatology. To this end, an adequate energy and protein intake will be ensured and the consumption of plant-based foods will be promoted to ensure an adequate intake of vitamins, minerals and antioxidants
  Arms: Intervention group
Behavioral: Physical exercise intervention — Weekly physical exercise guidelines will be given following the published Canadian clinical guideline recommendations combining moderate and vigorous aerobic activity. Walking will be performed 3 days a week for 30 minutes at a modified Borg scale intensity of 4-5/10, and 2 days a week for 15 minutes at a modified Borg scale intensity of 7-8/10. There will also be 5 minutes of warm-up and 5 minutes of recovery, in moderate activity at 3/10, and in vigorous activity at 4/10. In addition, 3 days per week (not coinciding with vigorous aerobic activity) of strength training at a modified Borg scale intensity of 7/10 will be included. Two sets of 8-10 repetitions will be performed, adaptable to that intensity according to the progression of the subjec
  Arms: Intervention group

SUMMARY:
The main aim of this study is to determine the effect of a multimodal intervention (Nutrition and Exercise) on quality of life, emotional well-being, and secondary symptomatology in patients diagnosed with breast cancer during neoadjuvant chemotherapy treatment, and to compare them with the control group.

DETAILED DESCRIPTION:
Multiple studies have demonstrated the relationship between obesity, sedentary lifestyle and stress on the risk of developing various types of cancer, including breast cancer. The correlation between a high Body Mass Index (BMI) and a worse prognosis in patients already diagnosed with breast cancer has also been studied, as well as the tendency to gain weight during chemotherapy treatments. A low-fat dietary pattern has been associated with reduced mortality after a breast cancer diagnosis, through mechanisms that decrease the likelihood of developing metabolic syndrome and reduce estradiol levels. In recent years, the importance of healthy lifestyle habits in improving the quality of life of these patients has also been demonstrated.

Although BMI is an easy-to-obtain marker of obesity, it is a rather crude measure that does not fully reflect the dysfunctional activity of visceral fat (VAT), which appears to be a key pathophysiological mechanism determining the clinical and metabolic consequences of obesity. Recent studies demonstrate an association between increased metabolic activity of VAT, determined preoperatively by 18F-FDG PET/CT, with the presence of metastatic axillary lymph node involvement in postmenopausal patients with luminal breast cancer.

The current study is proposed during neoadjuvant treatment (NY), and aims to determine whether after an intervention in exercise and diet improves the quality of life of patients and tolerability to oncological treatment NY. In addition, the investigators will use 18F-FDG PET/CT as a marker of aggressiveness at diagnosis by quantifying the metabolic activity of VAT (SUVmax VAT, SULmax VAT and VAT/SAT ratio) and subsequently in the assessment of response to treatment. The investigators will also determine the response at the histopathological level of the tumor itself after the intervention (residual tumor burden (RCB), Ki 67, TNM) and at the level of inflammation-related parameters (TNF, IL6, CRP), which can influence the prognosis and the risk of local or distant recurrence in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer who will undergo neoadjuvant treatment in the Oncology Unit of the Virgen de las Nieves University Hospital of Granada.
* Aged between 18 and 75 years.
* Give their consent to participate in the study and commit to complete the entire intervention and attend their follow-up appointments.
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols

Exclusion Criteria:

* Patients who are unwilling or unable to comply with the established guidelines by means of an intervention in diet and physical exercise and/or who present physical or psychological pathologies that contraindicate their inclusion in the study.
* Patients who do not register the data required for follow-up.
* Any condition that, in the investigator's opinion, impairs the ability to participate in the study or represents a personal risk for the participant.
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Participant's quality of life | 6 months
  QLQ-CD30 test
Participant's quality of life | 6 months
  BR23 test
Body composition | 6 months
  Weight (kg)
Body composition | 6 months
  Height (cm)
Body composition | 6 months
  Circumferences (waist and hip; cm)
Body composition | 6 months
  Fat mass (kg), visceral fat (g), lean mass (kg) and bone mineral content (g) will be evaluated by Dual Energy X-Ray Absorptiometry (Discovery Wi, Hologic Bedford, MA, USA) and 18F-FDG PET/CT

SECONDARY OUTCOMES:
Response rate | 6 months
  Response rate (%) determined by magnetic Resonance Imaging (MRI) and 18F-FDG PET/CT
Analytical parameters | 6 months
  Inflammation parameters: to analyze the degree of inflammation the modified Glasgow Pronostic Score (mGPS) is used, which is nowadays considered an important predictive tool for morbidity and mortality in these patients by measuring serum albumin and CRP values. IL6 and TNF levels, measured in pg/ml, which will be determined in blood samples.
Analytical parameters | 6 months
  Biochemical parameters: A routine analysis will be carried out in the Granada Hospital complex to determine biochemical parameters.
Analytical parameters | 6 months
  Biochemical parameters: A routine analysis will be carried out in the Granada Hospital complex to determine tumor markers.
Physical parameters | 6 months
  Muscle strength: By means of the manual grip test, completing two repetitions with each hand, with one minute between repetitions. A Takei 5401 Grip-D digital manual dynamometer (Takei, Tokyo, Japan) will be used.
Physical parameters | 6 months
  PAR-7 survey (to evaluate the previous physical level of the patients, it will be carried out via telephone by a single interviewer for all the patients included)
Emotional wellbeing | 6 months
  Beck Depression Inventory (BDI-II). Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe
Nutritional assessment | 6 months
  food frequency questionnaire which will asess the consumption of different food groups and nutrients intake.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas J Jurado-Fasoli, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided